CLINICAL TRIAL: NCT03482531
Title: Assessing, Depending on Personalized Manner, a Predicted Time to Delivery in the Context of Cervical Ripening With Dinoprostone Vaginal Insert
Brief Title: Assessing a Predicted Time to Delivery in the Context of Cervical Ripening With Dinoprostone Vaginal Insert
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: PHRC 2018-03
Record Dates: First submitted 2018-03-08; First posted 2018-03-29 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Dinoprostone Vaginal Insert
Keywords: limit nocturnal activity; cervical ripening
MeSH Terms: interventions — Models, Theoretical

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- before group: In the "before" group, the investigators retrospectively included 405 patients who had a dinoprostone vaginal insert for cervical ripening before induction of labor, between January 2015 and September 2016.
  Multivariate and regression analysis showed that the factors significantly increasing the time to delivery were: Nulliparity, obesity, a closed cervix on initial examination, and intact membranes at the time of insertion. The investigators also described a regression equation that allows to calculate the mean time from insert placement to delivery for each patient.
- after group: The investigators will prospectively include all eligible patients with a vaginal dinoprostone insert for cervical ripening during the next two years, starting on April 1st, 2018. At Angers hospital, there are around 600 cases of dinoprostone vaginal inserts per year, so the investigators will be able to include 400 to 500 patients during the study's duration.
  The equation will be incorporated when scheduling patients for cervical ripening with vaginal dinoprostone insert. The main objective of this study is to analyze to evaluate our mathematical model. One of the secondary objectives is to analyze whether the use of the personalized scheduling based on the mathematical model would decrease the rate of nocturnal deliveries (between midnight and 6 a.m.).
  Interventions: Other: mathematical model

INTERVENTIONS:
Other: mathematical model — mathematical model: regression equation that calculates the mean time from insert placement to delivery for each patient, based on every patient's characteristics (parity, BMI, cervical dilation and state of membranes)
  Groups: after group

SUMMARY:
Induction of labor is a common obstetric procedure that is routinely performed worldwide. However, when cervical conditions are not favorable (bishop <6), induction of labor is preceded by cervical ripening, usually with prostaglandins. The method of ripening most commonly used in France (89% of maternity wards) is the dinoprostone vaginal insert. In the majority of hospitals in France, dinoprostone vaginal inserts are usually placed in the morning, because of the higher availability of personnel (midwives and nurses). However, morning placement might increase the likelihood of the delivery occurring at night, since the mean interval between the insert placement and delivery is about 13 to 20 hours. Many studies have now shown that the risk of obstetrical complications, as well as neonatal morbidity and mortality is increased when deliveries occur at night. Several factors have been suggested behind the increased morbidity at night, including the lower number of personnel working, the fatigue associated with night work and the disruption of the circadian rhythm, and the insufficient supervision of residents.

Very few studies have evaluated the importance of the timing of placement of the intravaginal dinoprostone insert, and its influence on the occurrence of night deliveries. Some investigators have recently performed a retrospective study at Angers university hospital that assessed the time interval between placing the dinoprostone vaginal insert and delivery, as well as the factors impacting the time to delivery, and found that nulliparity, obesity, a closed cervix on initial examination, and intact membranes at the time of insertion increased the time to delivery. Moreover, the investigators proposed a regression equation that allows to calculate the mean time from insert placement to delivery for each patient, and have decided to incorporate it in the routine practice.

The investigators have decided to analyze the validity of the mathematical model. The consequence would be, thanks to a personalized timing for placement of dinoprostone vaginal insert based on every patient's characteristics (parity, BMI, cervical dilation and state of membranes), a decreased number of deliveries occurring between 12 p.m. and 6 a.m.

DETAILED DESCRIPTION:
This is a before-after, retrospective and prospective monocentric study. Patients in the "before" group were part of another study which are currently in the process of publishing and were retrospectively included, whereas patients in the "after" group will be prospectively included.

In the "before" group, the investigators retrospectively included 405 patients who had a dinoprostone vaginal insert for cervical ripening before induction of labor, between January 2015 and September 2016. The main outcome of the previous study was to evaluate the time interval between placing the dinoprostone vaginal insert and delivery. One of the secondary objectives was to determine the factors that would impact the time to delivery. Multivariate and regression analysis showed that the factors significantly increasing the time to delivery were: Nulliparity, obesity, a closed cervix on initial examination, and intact membranes at the time of insertion. The investigators also described a regression equation that allows to calculate the mean time from insert placement to delivery for each patient:

Y = 961,188 - 80,346 x parity + 21,437 x Body Mass Index (BMI) - 165,263 x cervical dilation- 241,759 x Premature rupture of membranes.

Following this study, the investigators decided to modify the routine procedures on the maternity ward and incorporate the equation when scheduling patients for cervical ripening with vaginal dinoprostone insert. The aim is to have a more personalized insertion schedule that would lower the number of deliveries occurring between midnight and 6 a.m., since it has been proven that there is a higher risk of obstetrical morbidity with night-time labor and delivery.

The investigators will prospectively include all eligible patients with a vaginal dinoprostone insert for cervical ripening during the next two years, starting on April 1st, 2018. At Angers hospital, there are around 600 cases of dinoprostone vaginal inserts per year, so 400 to 500 patients will be included during the study's duration. The investigators will then compare the outcomes in these patients that will comprise the "after" group, to the outcomes of patients in the "before" group, who delivered before the implementation of the new scheduling process. The investigators will thus be able to able to assess whether the mathematical model they suggested to estimate time to delivery and the personalized insertion timings have been confirmed. Then, subsequently, the objective is to analyze whether the use of the personalized scheduling based on the mathematical model they described would decrease the rate of nocturnal deliveries (between midnight and 6 a.m.).

The research project has been approved by the ethics committee of Angers university hospital on January 31st, 2018.

ELIGIBILITY:
Inclusion Criteria:

* have cervical ripening with the dinoprostone vaginal insert
* 34 weeks gestational age (GA) and beyond
* singleton pregnancies
* cephalic presentations

Exclusion Criteria:

* term < 34 weeks GA
* previous history of cesarean section
* women who refuse to participate in the study or have their data used.
* twin pregnancy
* prostaglandin allergies

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All eligible patients with a vaginal dinoprostone insert for cervical ripening ( because of not favorable cervical conditions (bishop <6) and needing induction of labor)
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-11-01 (Estimated); Study Completion 2019-11-01 (Estimated)

PRIMARY OUTCOMES:
Difference (in minutes) between the actual time to delivery compared to the predicted time | 2 days
  there will be different categories:
  * less than 180 minutes
  * more than 180 but less than 360 minutes
  * more than 360 but less than 540 minutes
  * more than 540 but less than 720 minutes
  * more than 720 minutes

SECONDARY OUTCOMES:
rate of deliveries | 2 years
  rate of deliveries occurring between midnight and 6 a.m. following cervical ripening with dinoprostone vaginal insert.
the Apgar score | 1, 3 and 5 minutes after delivery
  Apgar score lower than 7 at 1, 3 and 5 minutes. Apgar score lower than 7 at 5 minutes is correlated on the immediate child's development
neonatal potential of hydrogen (pH) | 1 hour
  * mean of neonatal potential of hydrogen (pH)
  * potential of hydrogen < 7.20 means foetal acidosis
  * potential of hydrogen is measured in the artery of umbilical cordon few minutes after delivery
  * potential of hydrogen lower than 7 leads to foetal acidosis responsible for neonatal encephalopathy
neonatal intensive care hospitalization | 12 hours
  The rate of neonatal intensive care hospitalization in the immediate postpartum and during the 12 hours after delivery
post-partum bleeding | 24 hours
  * the rate of post-partum bleeding
  * postpartum hemorrhage is a bleeding more than 500ml
  * severe postpartum hemorrhage is a bleeding more than 1000ml
Operative deliveries | 2 years
  the rate of forceps deliveries and vacuum extractions during the study duration
Cesarean sections | 2 years
  the rate of cesarean sections during the study duration

CONTACTS AND LOCATIONS:
Locations (1):
- Angers University hospital, Angers, Maine Et Loire, France

IPD SHARING:
Plan to Share IPD: Undecided